CLINICAL TRIAL: NCT06303791
Title: Digital-based Psychosocial Intervention for Parents of Children With Neurodevelopmental Disorders: a Randomized Control Trial
Brief Title: Digital-based Psychosocial Intervention for Parents of Children With Neurodevelopmental Disorders
Acronym: INPSYD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Carmen Berenguer-Forner, Profesor Permanent Lecturer - Department of Developmental and Educational Psychology, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1905517
Record Dates: First submitted 2024-03-04; First posted 2024-03-12 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Autism Spectrum Disorder; Attention Deficit Hyper Activity
Keywords: Psychosocial program; Autism; ADHD; RCT
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder; Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: To test the proposed objectives, a design will be used with a between-groups factor (type of therapy) and a intra-groups with pre-treatment (T0), post-treatment (T1) and follow-up measurements at 6 months (T2). Participants will be randomly assigned (1:1) to the two conditions; a group that will receive the intervention of the structured psychosocial program with digital support (experimental group) and an active control group. The experimental group will undergo an evaluation prior to the intervention, one immediately after it, and a third follow-up evaluation. In the case of the control group, it will be evaluated through the pretest phases, posttest and follow-up.
Who Masked: Participant, Outcomes Assessor
Masking Description: Families/children who meet the inclusion criteria will be randomly assigned to one of the two conditions (intervention group or control group) using a controlled design. Block randomization will be applied to each of the diagnostic groups (ASD, ADHD) to ensure that participants were of approximately similar size (1:1 ratio) in the treatment and control conditions. After determining the size of each block in the sample (#ASD and #ADHD) the treatment allocation of each individual participant will be done randomly.A blind procedure will be used: participating families will not know the group to which participants will be assigned, and the researchers who will collect and enter the data will also have no knowledge of the condition to which the families will be assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital Psychosocial Intervention group (Experimental): The intervention group will be made up of five successive groups of 8 to 10 families that will receive 12 weekly 90-minute sessions in a synchronous virtual mode by zoom platform The integrity of the sessions will be guaranteed by a digital manual that clearly outlined all the procedures to be used in the intervention. Additionally, sessions will be audiotaped and reviewed by a team member through a checklist to ensure groups receive equivalent set of information.
  Interventions: Behavioral: Digital Psychosocial intervention
- Control group (No Intervention): The control group of parents will be made up of another five successive groups of 8 to 10 families who will receive 12 sessions weekly 90 minutes. In these sessions these families will be encouraged to discuss their thoughts and share their experiences in a non-directive environment. The therapist will not be allowed to provide specific psychotherapy, psychoeducation or psychosocial techniques, nor any additional comments or information, but rather to guide the groups and allow everyone to express and give their personal point of view. The use of an active control group will ensure that the observed benefits are primarily due to the digitally supported psychosocial program only.

INTERVENTIONS:
Behavioral: Digital Psychosocial intervention — The psychosocial program with digital support has been developed by combining different theoretical perspectives on intervention in children with ASD without intellectual disabilities and children with ADHD. The contents of the program are based on three main approaches, each of which has separately demonstrated evidence in the treatment of these neurodevelopmental disorders: psychoeducation and stress management, cognitive behavioral techniques, and techniques in social and communication skills (Dahl et al., 2020; DuPaul et al., 2020; Tan-MacNeill et al., 2021).
  Arms: Digital Psychosocial Intervention group

SUMMARY:
The goal of this clinical trial is to implement a structured psychosocial intervention program with digital support (randomized and with a control group) that will be conducted virtually and synchronously to families of children with autism spectrum disorder (ASD) and families of children with Attention Deficit with hyperactivity Disorder (ADHD). The main questions it aims to answer are:

1. Will the program impact on different variables in the parents' domain (parental stress variables, quality of life/social support and coping skills),
2. Will the program impact on different variables in the children's domain (daily life functioning, social behavioral variables, and executive functioning).
3. Treatment outcomes will be assessed at pre-test, post-test, and 6-month follow-up assessment across intervention and control groups using a battery of measures of parenting stress, coping skills, social support, and children's dysfunctional outcomes

Parents and teachers will complete different questionnaires to see if there are improvements on parent's and children outcomes.

Researchers will compare intervention group and control group to see if there are improvements on parent's domains (parenting stress, coping skills, social support) and children's dysfunctional outcomes (daily life functioning, social behavioral variables, and executive functioning).

DETAILED DESCRIPTION:
AIMS The goal of this clinical trial is to implement a structured psychosocial intervention program with digital support (randomized and with a control group) that will be conducted virtually and synchronously to families of children with autism spectrum disorder (ASD) and families of children with Attention Deficit with hyperactivity Disorder (ADHD).

The specific aims of this study are:

1. to analyze whether a digital-based psychosocial program for parents of children with ASD and children with ADHD leads to an improvement of parent's outcomes (level of stress, coping skills, and perceived social support), in comparison with an active control group
2. to examine whether a digital-based psychosocial program for parents of children with ASD and children with ADHD will lead to improvement of children outcomes, such as social difficulties, daily executive disfunctions, and sleep or learning problems, in comparison with an active control group
3. Treatment outcomes will be assessed at pre-test, post-test, and 6-month follow-up assessment across intervention and control groups using a battery of measures of parenting stress, coping skills, social support, and children's dysfunctional outcomes

METHODOLOGY

Design

The basic research design is a randomized controlled design observing the recommendations made by Jadad and Enkin (2007). To test the proposed objectives, a mixed design will be used with a between-groups factor (type of therapy) and a intra-groups with pre-treatment (T0), post-treatment (T1) and follow-up measurements at 6 months (T2). Participants will be randomly assigned (1:1) to the two conditions; a group that will receive the intervention of the structured psychosocial program with digital support (experimental group) and a control group. The experimental group will undergo an evaluation prior to the intervention, one immediately after it, and a third follow-up evaluation. In the case of the control group, it will be evaluated through the pretest phases, posttest and follow-up.

Participants:

The present study enrolled 90 families of boys and girls with ASD without intellectual disabilities and ADHD, with an age range between 7 and 11 years (47 children with ASD without intellectual disabilities, and 43 children with ADHD). The children were recruited from specialized psychoeducational centers and medical centers in Spain. Informed consent will be requested from parents.

Sample size was calculated using a priori Sample Size Calculator for one-way ANOVA using G*power v. 3.1.9.4 setting the size of Type I error (significance level) of 0.05 (a) and the power of the study of the 80 %, anticipating an effect size (Cohen d) of 0.8.

Instruments:

Parents and teachers will complete different questionnaires to see if there are improvements on parent's domains and children's dysfunctional outcomes.

Researchers will compare intervention group and control group to see if there are improvements on parent's domains and children's dysfunctional outcomes

Procedure:

The study was approved by the Ethics Committee of the Universitat de València in accordance with the principles of Helsinki Declaration (World Medical Association,2013) (UV-INV_ETICA-1,905,517). The tests were applied by psychologists who were familiar with the use of the different instruments. The parents provided their written informed consent, in addition to the oral consent of all the children who participated This study was supported by the Spanish project PID2021-128044NA-100 (Ministerio de Ciencia e Innovacion/AEI/FEDER, UE)

Families/children who meet the inclusion criteria will be randomly assigned to one of the two conditions (intervention group or control group) using a controlled design. Block randomization will be applied to each of the diagnostic groups (ASD, ADHD) to ensure that the participants were of approximately similar size (1:1 ratio) in the treatment and control conditions. After determining the size of each block in the sample (#ASD and #ADHD) the treatment allocation of each individual participant will be done randomly.A blind procedure will be used: participating families will not know the group to which the participants will be assigned, and the researchers who will collect and enter the data will also have no knowledge of the condition to which the families will be assigned.

The intervention program, as well as the evaluation, will be carried out by an expert psychologist in neurodevelopmental disorders. The psychosocial program with digital support has been developed by combining different theoretical perspectives on intervention in children with ASD without intellectual disabilities and children with ADHD. The contents of the program are based on three main approaches, each of which has separately demonstrated evidence in the treatment of these neurodevelopmental disorders: psychoeducation and stress management, cognitive behavioral techniques, and techniques in social and communication skills (Dahl et al., 2020; DuPaul et al., 2020; Tan-MacNeill et al., 2021).

The intervention sessions with parents will be carried out in a synchronous virtual mode with the aim of achieving maximum adherence to the program and overcoming logistical barriers of physical distances, and the problems of coping with work and care. The sessions will be in small groups to adapt to these needs. Specifically, the psychosocial intervention group will be made up of five successive groups of 8 to 10 families that will receive 12 weekly 90-minute sessions.

The integrity of the sessions will be guaranteed by a digital manual that clearly outlined all the procedures to be used in the intervention. Additionally, sessions will be audiotaped and reviewed by a team member through a checklist to ensure groups receive equivalent set of information.

The control group of parents will be made up of another five successive groups of 8 to 10 families who will receive 12 sessions weekly 90 minutes. In these sessions these families will be encouraged to discuss their thoughts and share their experiences in a non-directive environment. The therapist will not be allowed to provide specific psychotherapy, psychoeducation or psychosocial techniques, nor any additional comments or information, but rather to guide the groups and allow everyone to express and give their personal point of view. The use of an active control group will ensure that the observed benefits are primarily due to the digitally supported psychosocial program only.

Both groups will have the same conditions at baseline and the sessions will be carried out by the same therapist in both groups. Likewise, another person from the research team will verify the integrity of the program.

The pre- and post-test evaluation of the parents will be carried out in person individually in a meeting room of the Faculty of Psychology of University of Valencia. Likewise, before the first intervention session, parents will be provided with a tutorial on the video conferencing platform (Zoom, <www.zoom.us>) to familiarize with the software and minimize potential risks. Parents will be able to participate in the program from home or another location, as long as parents have an internet connection, using a tablet, computer or smartphone, with a webcam. Zoom has been chosen because it can host online group meetings without an annual commitment, unlike other types of software. Zoom is has been used successfully in health research. Participants can access meetings without having to purchase or install software through any device. Participants will be able to access the meetings online through a hyperlink, or log in the ID and password that will be provided to the participants and to enter the session.

Continuous contact will be maintained via telephone and virtual with families, to provide an immediate response to any difficulty that may arise in the intervention process.

The Structure of a typical session: (90mn) in experimental group would be:

* Welcome / questions doubts previous session
* Theoretical explanation on the topic of the session
* Modeling and roll-playing, videos on the contents explained (e.g. cognitive techniques and/or relaxation techniques)
* Proposal of activities for the week based on the contents explained in each session
* Questionnaire of questions about content and satisfaction with the session

Plan for missing data:

The investigators will use different statistical methods to deal with missing data, specifically participants with any missing data will be excluded from analysis or the investigators will use a simple mean imputation being very cautious not to bias the method

Statistical analysis:

Statistical analyzes will be carried out based on the objectives set, trying to control the contaminating effects as much as possible.

Preliminary analyzes will be carried out (Kolmogorov-Smirnov test) to confirm the assumptions of normality maintained between the different variables. Non-parametric or parametric tests will be applied, depending on whether the criteria to perform the tests are met.

For intragroup comparisons, repeated measures ANOVAs will be run to evaluate the change in the pre/posttest results and in the follow-up six months later. Descriptive statistics will be calculated, and other statistics will be applied (e.g. Mann-Whitney U statistic) for comparison between experimental groups, performing moderation analysis with the conceptually indicated variables. Effect sizes will be calculated using partial eta squared values (according to Cohen (1988) an eta squared, 0.06 = small; 0.06-0.14 = medium; 0.14 = large). Statistical analyzes will be carried out with the SPSS v statistical package. 24.0.

ELIGIBILITY:
Inclusion Criteria:

* 1) diagnosis of ASD according to Autistic Diagnostic Interview-Revised (ADI-R; Rutter at al., 2006), and/or the Autism Diagnostic Observation Schedule, Generic (ADOS G; Lord et al., 2000) confirmed by child psychologist or ADHD any presentation according to the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition DSM-V; APA, (2013)] for parents and teachers
* 2) IQ> 80
* 3) age of children between 7 and 11 years, either sex
* 4) informed consent of the parents and the children available
* 5) parents' age greater than or equal to 18 years
* 6) responsibility and legal capacity in parents and access to internet.

Exclusion Criteria:

* Exclusion criteria included subjects with any medical or psychiatric condition, an IQ of less than 80, motor or sensorial deficits, and children whose families had received any psychosocial treatment before.

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2022-09-07 (Actual); Primary Completion 2024-11-17 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Parental stress in The Parenting Stress Index - Short Form (PSI-SF) Spanish adaptation | Baseline and week 12 and week 36
  The parental distress subscale is a validated parent questionnaire that measures the level of distress a parent experiences due to personal factors. The scale provides a measure of total stress by adding up the scores on the 36 items, with a total score above 90 being clinically significant. The PSI-SF presents good psychometric properties
Social support: The Social Functional Support Questionnaire Duke-UNC | Baseline and week 12 and week 36
  The Social Functional Support is a validated parent report Questionnaire that measures the subjects' perception of the availability of help from family and friends in difficult situations. The instrument comprises 11 questions with a Likert-type scale ranging from 1 = "much less than I would like" to 5 = "as much as I would like". Scores of less than 32 indicate low perceived social support. The questionnaire presents good psychometric properties
Coping Skills using The Brief COPE | Baseline and week 12 and week 36
  The Brief COPE is a validated parent questionnaire that measures the usage frequencies of broad-based maladaptive and adaptive coping strategies. Items are rated on a four-point rating scale ranging from 1= 'I haven't been doing this at all' to 4= 'I've been doing this a lot'. The psychometric properties of the Brief COPE are good
Children's social problems using Strengths and Difficulties Questionnaire (SDQ) | Baseline and week 12 and week 36
  The SDQ is a validated parent report questionnaire. This questionnaire has 25 items and is designed for children from 4 to 16 years old. The items are divided into 5 subscales: Emotional symptoms, Behavioral problems, Hyperactivity, Peer relationship problems, and Prosocial behaviors. In addition, it has a total difficulty score of behavioral problems obtained by adding together all the subscales except prosocial behavior. The items are scored on a Likert-type scale from 1 (not true) to 3 (completely true). On all the scales, a higher score implies greater difficulty, except the prosocial behavior scale, where a higher score is more positive than a lower one. The questionnaire presents good psychometric properties
Daily life executive functioning using the BRIEF | Baseline and week 12 and week 36
  The Behavioral Rating Inventory of Executive Function (BRIEF-2 Family report is a questionnaire completed by a relative/caregiver, which assesses daily executive functions. It consists of 63 items that are answered on a frequency scale (never, sometimes, and frequently). The raw scores are transformed into age-corrected T-scores. A score greater than 70 on any of the scales indicates clinically significant difficulties. Very high internal consistency has been reported

SECONDARY OUTCOMES:
Children Sleep problems: using The Sleep Disturbance Scale for Children (SDSC) | Baseline and week 12 and week 36
  The Sleep Disturbance Scale for Children s a 26-item parent-reported questionnaire that assesses the occurrence of sleep disturbances during the last 6 months in children aged 6-16 years. The 26 items are rated on a 5-point scale (never to always), yielding a continuous variable ranging from 26 to 130 with higher values reflecting a greater severity of symptoms. The instrument has good psychometric properties
Behavioral problems using The Weiss Functional Impairment Rating Scale-Parent Form (WFIRS-P) | Baseline and week 12 and week 36
  The Weiss Functional Impairment Rating Scale-Parent Form (WFIRS-P) is a 50-item scale that requires parents to rate the impact of their child's emotional or behavioural problems in the previous month on six separate domains: family, school and learning; life skills; child's self-concept; social activities; and risky activities. Each item is rated on a four-point scale from 0 ('never or not at all') to 3 ('very often or very much') or as 'not applicable'. Higher scores indicate behavioral difficulties. Raw scores are used. The questionnaire has good psychometric properties
Children Learning Behavior using Learning behavior scale (LBS) | Baseline and week 12 and week 36
  The LBS is a validated teacher questionnaire that measures student behaviors related to effective and efficient learning. The Learning Behaviors Scale contains 29 items, six items with positive wording and the remaining items with relatively negative wording in order to reduce response sets. Items are rated on a 3-point Likert scale (0 D Does not apply, 1 D Sometimes applies, 2 D Most often applies). High scores indicate good learning behavior, and low scores are interpreted as faulty learning behavior. The instrument has good psychometric properties

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Berenguer, PhD, Principal Investigator — University of Valencia
Locations (1):
- University of Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Immediately following publication. No end date.
Access Criteria: Anyone who wishes to access the data.
URL: https://roderic.uv.es/home

REFERENCES:
- [Background] Davis NO, Kollins SH. Treatment for co-occurring attention deficit/hyperactivity disorder and autism spectrum disorder. Neurotherapeutics. 2012 Jul;9(3):518-30. doi: 10.1007/s13311-012-0126-9. PMID 22678458
- [Background] Young S, Hollingdale J, Absoud M, Bolton P, Branney P, Colley W, Craze E, Dave M, Deeley Q, Farrag E, Gudjonsson G, Hill P, Liang HL, Murphy C, Mackintosh P, Murin M, O'Regan F, Ougrin D, Rios P, Stover N, Taylor E, Woodhouse E. Guidance for identification and treatment of individuals with attention deficit/hyperactivity disorder and autism spectrum disorder based upon expert consensus. BMC Med. 2020 May 25;18(1):146. doi: 10.1186/s12916-020-01585-y. PMID 32448170
- [Background] van Steijn DJ, Oerlemans AM, van Aken MA, Buitelaar JK, Rommelse NN. The reciprocal relationship of ASD, ADHD, depressive symptoms and stress in parents of children with ASD and/or ADHD. J Autism Dev Disord. 2014 May;44(5):1064-76. doi: 10.1007/s10803-013-1958-9. PMID 24114582
- [Background] Craig F, Operto FF, De Giacomo A, Margari L, Frolli A, Conson M, Ivagnes S, Monaco M, Margari F. Parenting stress among parents of children with Neurodevelopmental Disorders. Psychiatry Res. 2016 Aug 30;242:121-129. doi: 10.1016/j.psychres.2016.05.016. Epub 2016 Jun 1. PMID 27280521
- [Background] Siegenthaler-Hierro R, Presentacion-Herrero MJ, Colomer-Diago C, Miranda-Casas A. [Moderators of psychosocial intervention in preschoolers with attention deficit hyperactivity disorder]. Rev Neurol. 2013 Feb 22;56 Suppl 1:S85-92. Spanish. PMID 23446728
- [Result] DuPaul GJ, Evans SW, Mautone JA, Owens JS, Power TJ. Future Directions for Psychosocial Interventions for Children and Adolescents with ADHD. J Clin Child Adolesc Psychol. 2020 Jan-Feb;49(1):134-145. doi: 10.1080/15374416.2019.1689825. Epub 2019 Dec 4. PMID 31799864
- [Result] Montoya A, Colom F, Ferrin M. Is psychoeducation for parents and teachers of children and adolescents with ADHD efficacious? A systematic literature review. Eur Psychiatry. 2011 Apr;26(3):166-75. doi: 10.1016/j.eurpsy.2010.10.005. Epub 2011 Feb 2. PMID 21292454
- [Result] Ferrin M, Moreno-Granados JM, Salcedo-Marin MD, Ruiz-Veguilla M, Perez-Ayala V, Taylor E. Evaluation of a psychoeducation programme for parents of children and adolescents with ADHD: immediate and long-term effects using a blind randomized controlled trial. Eur Child Adolesc Psychiatry. 2014 Aug;23(8):637-47. doi: 10.1007/s00787-013-0494-7. Epub 2013 Dec 1. PMID 24292412
- [Result] Tan-McNeill, K. M., Smith, I. M., Johnson, S. A., Chorney, J., & Corkum, P. (2021). A systematic review of online parent-implemented interventions for children with neurodevelopmental disorders. Children's Health Care, 1-39.
- [Result] Sonuga-Barke EJ, Daley D, Thompson M, Laver-Bradbury C, Weeks A. Parent-based therapies for preschool attention-deficit/hyperactivity disorder: a randomized, controlled trial with a community sample. J Am Acad Child Adolesc Psychiatry. 2001 Apr;40(4):402-8. doi: 10.1097/00004583-200104000-00008. PMID 11314565
- [Result] Sadeghi S, Pouretemad HR, Shalani B. Internet-based versus face-to-face intervention training for parents of young children with excessive screen-time and autism spectrum disorder-like symptoms: a comparative study. Int J Dev Disabil. 2021 Mar 8;68(5):744-755. doi: 10.1080/20473869.2021.1895699. eCollection 2022. PMID 36210895
- [Derived] Pardo-Salamanca A, Gomez S, Santamarina C, Pastor G, Berenguer C. The effectiveness of an online-based psychosocial program for parents of children with neurodevelopmental disorders - a randomized controlled trial. Child Adolesc Ment Health. 2025 Nov 5. doi: 10.1111/camh.70044. Online ahead of print. PMID 41193165